CLINICAL TRIAL: NCT02369835
Title: A Randomized Study of Topical Dilute Hypochlorite (Modified Dakin's Solution) Treatment for the Prevention of Radiation Dermatitis in Head and Neck Cancer
Brief Title: Modified Dakin's Solution in Reducing Radiation-Induced Dermatitis in Patients With Head and Neck Cancer Undergoing Radiation Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Beth Beadle, Associate Professor of Radiation Oncology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: IRB-32439; NCI-2015-00176 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB-32439 (Other: Stanford IRB); ENT0042 (Other: OnCore)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Results first posted 2019-09-17 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Head and Neck Carcinoma; Radiation-Induced Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Sodium Hypochlorite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (modified Dakin's solution) (Experimental): Participants apply modified Dakin's solution (0.005% to 0.010%) topically to the skin of the arm up to 3 hours in advance of each radiation treatment.
  Interventions: Drug: Dakin's solution
- Arm II (placebo) (Placebo Comparator): Participants apply placebo solution (saline) topically to the skin of the arm up to 3 hours in advance of each radiation treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dakin's solution — Apply modified Dakin's solution (0.005 to 0.01%) topically
  Other Names: Sodium hypochlorite in aqueous solution; Dakin's fluid; Liquid bleach
  Arms: Arm I (modified Dakin's solution)
Other: Placebo — Applied topically
  Other Names: PLCB
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase 3 trial studies how well modified Dakin's solution works in reducing radiation-induced dermatitis, a common skin reaction to radiation therapy, in patients with head and neck cancer undergoing radiation therapy. Modified Dakin's solution may reduce inflammation in the body, which may prevent or reduce dermatitis after radiation therapy.

Radiation therapy in this study is regulatory medical care based on the patient's needs and the radiation oncologist's judgment. It is not possible nor necessary to explicitly define the dose or duration of treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the proportion of patients who develop grade 3 radiation dermatitis (as defined by the Stanford Radiation Dermatitis Scoring System) as an adverse effect of radiation therapy or chemoradiation therapy for a head and neck cancer when initiating the use of prophylactic hypochlorite (HOCl) (modified Dakin's solution) at the start of therapy (experimental arm) compared to placebo (control arm).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (EXPERIMENTAL): Participants apply modified Dakin's solution (0.005% to 0.010%) topically to the skin of the arm up to 3 hours in advance of each radiation treatment.

ARM II (CONTROL): Participants apply placebo solution (saline) topically to the skin of the arm up to 3 hours in advance of each radiation treatment.

At the time that Stanford Radiation Dermatitis Scoring System (SRDSS) Grade E radiation dermatitis develops, the participant will transition to standard management for radiation dermatitis. SRDSS, by grade, is as follows.

* A. No skin change
* B. Faint, barely detectable erythema
* C. Follicular rash, hyperpigmentation, evolving erythema
* D. Dry desquamation, brisk erythema
* E. Moist desquamation
* F. Bleeding, ulceration, and/or infection

SRDSS Grade E is roughly equivalent to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 Grade 3 radiation dermatitis, "Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion."

After completion of study, patients are followed up at 6 to 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer who plan to undergo radiation therapy to the head and neck region
* At least 18 years of age
* Able to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Prior radiation therapy to the head and neck region or prior chemotherapy for head and neck cancer (induction chemotherapy NOT excluded)
* The physician-approved radiation treatment plan indicates a maximum prescription dose of less than 45 Gy
* Scleroderma or discoid lupus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-05; Primary Completion 2018-07-18 (Actual); Study Completion 2018-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Beadle, Principal Investigator — Stanford University Hospitals and Clinics
Locations (2):
- United States (2):
  - Stanford Cancer Center South Bay, San Jose, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Modified Dakin's Solution) | Arm II (Placebo)
Started | 64 | 68
Completed | 53 (Reasons that participants did not complete for the Primary Outcome are not available.) | 55 (Reasons that participants did not complete for the Primary Outcome are not available.)
Not Completed | 11 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Modified Dakin's Solution) | Arm II (Placebo) | Total
Number analyzed (Participants) | 64 | 68 | 132
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 42 | 71
  >=65 years | 35 | 26 | 61
Age, Continuous [Median (Standard Deviation); unit: years] | 66 (11.6) | 62 (12.7) | 63.5 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 14 | 24
  Male | 54 | 54 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 5 | 9 | 14
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 1 | 2 | 3
  White | 45 | 49 | 94
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 64 | 68 | 132
Baseline dermatitis [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Radiation Dermatitis
Description: Participants were assessed for radiation dermatitis on the arms according to the Stanford Radiation Dermatitis Scoring System (SRDSS), at baseline and through their treatment course. The outcome is reported by treatment group as the number and proportion of participants that experience SRDSS Grade E or greater radiation dermatitis through 10 weeks after completion of radiation treatment, a number without dispersion.
  SRDSS, by grade:
  * A. No skin change
  * B. Faint, barely detectable erythema
  * C. Follicular rash, hyperpigmentation, evolving erythema
  * D. Dry desquamation, brisk erythema
  * E. Moist desquamation
  * F. Bleeding, ulceration, and/or infection
  SRDSS Grade E is roughly equivalent to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 Grade 3 radiation dermatitis, "Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion"
Time Frame: From first radiation treatment up to 10 weeks after completion of radiation treatment. Because much of the study data was not provided by the prior investigator to the current Responsible Party, it is not possible to be more precise than stated.
Population: Not all participants completed radiation treatment, and are not included in the outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Modified Dakin's Solution) | Arm II (Placebo)
Number analyzed (Participants) | 53 | 55
Participants | 34 | 36
Statistical Analysis 1: Comparison: Arm I (Modified Dakin's Solution) vs Arm II (Placebo); Test type: Other; p = .8872, Chi-squared

2. Secondary Outcome: Time to Grade E Radiation Dermatitis
Description: Participants were assessed for radiation dermatitis on the arms according to the Stanford Radiation Dermatitis Scoring System (SRDSS), at baseline and through their treatment course. The time that SRDSS Grade E radiation dermatitis developed was noted. The outcome is reported by treatment group as the mean time to development of SRDSS Grade E radiation dermatitis, with standard deviation.
  SRDSS, by grade:
  * A. No skin change
  * B. Faint, barely detectable erythema
  * C. Follicular rash, hyperpigmentation, evolving erythema
  * D. Dry desquamation, brisk erythema
  * E. Moist desquamation
  * F. Bleeding, ulceration, and/or infection
  SRDSS Grade E is roughly equivalent to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 Grade 3 radiation dermatitis, "Moist desquamation in areas other than skin folds and creases; bleeding induced by minor trauma or abrasion."
  Additional information describing this outcome is not available.
Time Frame: up to 12 weeks (estimated)
Population: Data for time to Grade E radiation dermatitis was not provided by the prior investigator to the current Responsible Party. On this basis, data is not available, and will never be available.
Arm/Group | Arm I (Modified Dakin's Solution) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pain Associated With Radiation Dermatitis
Description: Quality of life was assessed as pain associated with radiation dermatitis. Assessments were baseline and through treatment follow-up 3 to 12 weeks after completion of radiation treatment. The assessment was to be conducted with a Modified Brief Pain Inventory (MBPI), a 13-question survey with responses ranging from 0 to 10, and an overall score of 0 to 130. A higher score indicates more pain and less quality of life. The outcome was to be reported by treatment group as the mean score with standard deviation.
  Additional information describing this outcome is not available.
Time Frame: 3 to 12 weeks after completion of radiation treatment
Population: Data for pain associated with radiation dermatitis was not provided by the prior investigator to the current Responsible Party. On this basis, data is not available, and will never be available.
Arm/Group | Arm I (Modified Dakin's Solution) | Arm II (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of the study - from consent to the end of follow-up (follow-up visit 3 to 12 weeks after completion of treatment). Because much of the study data was not provided by the prior investigator to the current Responsible Party, it is not possible to be more precise than stated.
Description: Reported adverse events represent the entire set of adverse events as available to the current investigator and Responsible Party. There are no additional events available to report, and there never will be.
Arm/Group | Arm I (Modified Dakin's Solution) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/68
Serious Adverse Events (participants affected / at risk) | 34/64 | 36/68
Other Adverse Events (participants affected / at risk) | 53/64 | 55/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Modified Dakin's Solution) (N=64) | Arm II (Placebo) (N=68)
Radiation dermatitis (Injury, poisoning and procedural complications) | 34 (34) | 36 (36)
Cardiac arrest (Cardiac disorders) | 1 (2) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Acneiform Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Other, Foot ulcer (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Other, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspiration, pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1)
Other, Feeding tube dysfunction (Surgical and medical procedures) | 0 (0) | 1 (1)
Pain, shoulder pain (General disorders) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Modified Dakin's Solution) (N=64) | Arm II (Placebo) (N=68)
Radiation dermatitis (Injury, poisoning and procedural complications) | 53 (53) | 55 (55) — Development of grade 1 or higher non-serious radiation dermatitis (per CTCAE)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/35/NCT02369835/Prot_SAP_001.pdf